CLINICAL TRIAL: NCT01457339
Title: A Phase 1, Randomized, Double-blind, Placebo Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ascending, Multiple Oral Doses of SPD489 (Lisdexamfetamine Dimesylate) in Clinically Stable Adults With Schizophrenia
Brief Title: Assess the Safety and Pharmacokinetics of Ascending, Multiple Oral Doses of SPD489 in Adults With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SPD489-119
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPD489 (Lisdexamfetamine dimesylate) (Experimental)
  Interventions: Drug: SPD489 (Lisdexamfetamine dimesylate)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 (Lisdexamfetamine dimesylate) — SPD489 administered orally in ascending doses (50mg, 70mg, 100mg, 150mg, 200mg, 250mg). Each of these doses will be administered once daily for 5 days. Total number of days dosed is 30 days.
  Other Names: Vyvanse, LDX
  Arms: SPD489 (Lisdexamfetamine dimesylate)
Drug: Placebo — Placebo Capsule(s) for oral use taken once daily for 30 days
  Arms: Placebo

SUMMARY:
This is a multiple ascending dose study; the purpose of this study is to examine the safety, tolerability and pharmacokinetics (levels of drug in the blood) of SPD489 in Schizophrenic Patients who are currently maintained on a stable dose of an antipsychotic medication.

ELIGIBILITY:
Subjects must be diagnosed with schizophrenia, on a stable dose of an antipsychotic and not have any cardiac risk factors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10-21 (Actual); Primary Completion 2012-01-20 (Actual); Study Completion 2012-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- United States (2):
  - California Clinical Trials, Glendale, California
  - Collaborative Neuroscience Network, Inc, Long Beach, California

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD489 (Lisdexamfetamine Dimesylate): Ascending multiple, oral doses of SPD489 (50mg, 70mg, 100mg, 150mg, 200mg, 250mg) administered once daily for 5 days at each dose level (30 days total).
Period: Period 1 (50 mg)
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)
Started | 7 | 24
Completed | 7 | 24
Not Completed | 0 | 0
Period: Period 2 (70 mg)
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)
Started | 7 | 24
Completed | 7 | 24
Not Completed | 0 | 0
Period: Period 3 (100 mg)
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)
Started | 7 | 24
Completed | 7 | 23
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 4 (150 mg)
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)
Started | 7 | 23
Completed | 7 | 23
Not Completed | 0 | 0
Period: Period 5 (200 mg)
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)
Started | 7 | 23
Completed | 7 | 22
Not Completed | 0 | 1
Not completed — Met stopping criteria for PANSS score | 0 | 1
Period: Period 6 (250 mg)
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)
Started | 7 | 22
Completed | 6 | 21
Not Completed | 1 | 1
Not completed — Family Emergency | 1 | 0
Not completed — Personal appointment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SPD489 (Lisdexamfetamine Dimesylate)(All Doses): Ascending multiple, oral doses of SPD489 (50mg, 70mg, 100mg, 150mg, 200mg, 250mg) administered once daily for 5 days at each dose level (30 days total).
- Total: Total of all reporting groups
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(All Doses) | Total
Number analyzed (Participants) | 7 | 24 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 24 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (4.93) | 46.4 (7.86) | 47.1 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 6 | 19 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 24 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Day 5: 50 mg
Description: Blood pressure and pulse measurements were taken using an automated blood pressure monitoring device (ideally using the same device, the same arm and in the same position throughout the study). Measurements of vital signs were performed in triplicate (3 measurements) after the subject had been in a sitting position for at least 5 minutes. Each of the 3 triplicate readings were performed in succession, at least 1-2 minutes apart, with the cuff fully deflated between measurements. It was expected that the triplicate measurements be obtained within a 5-6 minute period.
Time Frame: Baseline and day 5
Population: Safety Set consisted of subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo: Placebo Capsule(s) for oral use taken once daily for 5 days
- SPD489 (Lisdexamfetamine Dimesylate)(50 mg): Oral 50 mg dose of SPD489 administered once daily for 5 days.
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
mmHg | -0.14 (9.543) | 8.94 (11.510)

2. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Day 5: 70 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- SPD489 (Lisdexamfetamine Dimesylate)(70 mg): Oral 70 mg dose of SPD489 administered once daily for 5 days.
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
mmHg | 1.43 (12.593) | 3.82 (9.258)

3. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Day 5: 100 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- SPD489 (Lisdexamfetamine Dimesylate)(100 mg): Oral 100 mg dose of SPD489 administered once daily for 5 days.
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
mmHg | 0.43 (6.448) | 4.96 (9.208)

4. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Lisdexamfetamine Dimesylate on Day 5: 50 mg
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: Pharmacokinetic Set defined as all subjects in the Safety set who had evaluable concentration-time profiles for lisdexamfetamine and/or d-amphetamine.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 24
ng*hr/ml | 25.6 (12.9)

5. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Lisdexamfetamine Dimesylate on Day 5: 70 mg
Description: as for outcome 4
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 24
ng*hr/ml | 43.7 (27.5)

6. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Lisdexamfetamine Dimesylate on Day 5: 100 mg
Description: as for outcome 4
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 23
ng*hr/ml | 80.5 (37.2)

7. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Lisdexamfetamine Dimesylate on Day 5: 150 mg
Description: as for outcome 4
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Groups:
- SPD489 (Lisdexamfetamine Dimesylate)(150 mg): Oral 150 mg dose of SPD 489 administered once daily for 5 days.
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 22
ng*hr/ml | 144.9 (43.7)

8. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Lisdexamfetamine Dimesylate on Day 5: 200 mg
Description: as for outcome 4
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Groups:
- SPD489 (Lisdexamfetamine Dimesylate)(200 mg): Oral 200 mg dose of SPD489 administered once daily for 5 days.
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 21
ng*hr/ml | 230.2 (81.1)

9. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Lisdexamfetamine Dimesylate on Day 5: 250 mg
Description: as for outcome 4
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Groups:
- SPD489 (Lisdexamfetamine Dimesylate)(250 mg): Oral 250 mg dose of SPD489 administered once daily for 5 days.
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 21
ng*hr/ml | 301.5 (105.9)

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lisdexamfetamine Dimesylate on Day 5: 50 mg
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 24
ng/ml | 21.93 (9.96)

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lisdexamfetamine Dimesylate on Day 5: 70 mg
Description: as for outcome 10
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 24
ng/ml | 35.02 (21.35)

12. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Day 5: 150 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
mmHg | -2.81 (7.358) | 6.43 (13.519)

13. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Day 5: 200 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 23
mmHg | -2.38 (11.546) | 5.28 (11.761)

14. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Day 5: 250 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
mmHg | -0.28 (13.442) | 7.36 (15.569)

15. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Day 5: 50 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
mmHg | 2.86 (11.547) | 5.22 (8.364)

16. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Day 5: 70 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
mmHg | 2.38 (10.557) | 2.14 (6.468)

17. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Day 5: 100 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
mmHg | 2.14 (7.796) | 4.55 (7.641)

18. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Day 5: 150 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
mmHg | 2.67 (10.846) | 2.43 (10.672)

19. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Day 5: 200 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 23
mmHg | 2.76 (14.442) | 3.77 (8.041)

20. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Day 5: 250 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
mmHg | 3.67 (8.618) | 3.79 (10.106)

21. Primary Outcome: Change From Baseline in Pulse Rate at Day 5: 50 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
beats/min | 2.62 (9.534) | 3.78 (11.116)

22. Primary Outcome: Change From Baseline in Pulse Rate at Day 5: 70 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
beats/min | -0.95 (9.821) | 5.07 (9.500)

23. Primary Outcome: Change From Baseline in Pulse Rate at Day 5: 100 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
beats/min | 0.19 (10.306) | 5.72 (12.578)

24. Primary Outcome: Change From Baseline in Pulse Rate at Day 5: 150 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
beats/min | -1.05 (8.125) | 6.41 (13.782)

25. Primary Outcome: Change From Baseline in Pulse Rate at Day 5: 200 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 23
beats/min | 2.38 (10.058) | 8.88 (12.206)

26. Primary Outcome: Change From Baseline in Pulse Rate at Day 5: 250 mg
Description: as for outcome 1
Time Frame: Baseline and day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
beats/min | 2.06 (9.760) | 12.39 (12.666)

27. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lisdexamfetamine Dimesylate on Day 5: 100 mg
Description: as for outcome 10
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 23
ng/ml | 50.6 (18.9)

28. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lisdexamfetamine Dimesylate on Day 5: 150 mg
Description: as for outcome 10
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 22
ng/ml | 90.34 (30.45)

29. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lisdexamfetamine Dimesylate on Day 5: 200 mg
Description: as for outcome 10
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 21
ng/ml | 133.3 (63.17)

30. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lisdexamfetamine Dimesylate on Day 5: 250 mg
Description: as for outcome 10
Time Frame: Day 5 (12-hour sampling period post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 21
ng/ml | 181.53 (72.82)

31. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 5: 50 mg
Description: The PANSS is a validated measure that evaluates the presence, absence, and severity of 30 symptoms of schizophrenia including both positive and negative symptoms and general psychopathology. Each of the 30-items are rated on a scale of 1 (absent) to 7 (extreme) with a total scoring range of 30 to 210. Higher scores indicate more impairment.
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | 0.6 (2.22) | -1.9 (1.10)

32. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 5: 70 mg
Description: as for outcome 31
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | -2.1 (1.81) | -2.9 (1.50)

33. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 5: 100 mg
Description: as for outcome 31
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | -3.6 (1.43) | -3.9 (1.68)

34. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 5: 150 mg
Description: as for outcome 31
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | -2.1 (1.40) | -4.7 (1.44)

35. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 5: 200 mg
Description: as for outcome 31
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 22
units on a scale | -2.3 (2.01) | -4.6 (1.81)

36. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 5: 250 mg
Description: as for outcome 31
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
units on a scale | -2.3 (2.03) | -2.4 (2.01)

37. Secondary Outcome: Change From Baseline in Scale for the Assessment of Negative Symptoms (SANS-18) Total Score at Day 5: 50 mg
Description: The SANS was modified by eliminating the global and attention items; the score of the remaining non-global items is referred to as the SANS-18 total score. Each of the 18-items is scored on a scale from 0 (not at all) to 5 (severe) with a total scoring range of 0 to 90. Higher scores indicate more impairment.
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | -1.4 (1.54) | -1.7 (1.09)

38. Secondary Outcome: Change From Baseline in Scale for the Assessment of Negative Symptoms (SANS-18) Total Score at Day 5: 70 mg
Description: as for outcome 37
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | -3.0 (2.85) | -3.1 (1.15)

39. Secondary Outcome: Change From Baseline in Scale for the Assessment of Negative Symptoms (SANS-18) Total Score at Day 5: 100 mg
Description: as for outcome 37
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | -7.0 (3.07) | -2.6 (1.27)

40. Secondary Outcome: Change From Baseline in Scale for the Assessment of Negative Symptoms (SANS-18) Total Score at Day 5: 150 mg
Description: as for outcome 37
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | -4.0 (3.24) | -3.0 (1.17)

41. Secondary Outcome: Change From Baseline in Scale for the Assessment of Negative Symptoms (SANS-18) Total Score at Day 5: 200 mg
Description: as for outcome 37
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 22
units on a scale | 1.3 (3.75) | -2.6 (1.11)

42. Secondary Outcome: Change From Baseline in Scale for the Assessment of Negative Symptoms (SANS-18) Total Score at Day 5: 250 mg
Description: as for outcome 37
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
units on a scale | -4.2 (2.15) | -3.3 (1.47)

43. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Total Score at Day 5: 50 mg
Description: CDSS is a 9-item scale to evaluate depression in subjects who have schizophrenia rated from 0 (absence of symptoms) to 3 (severe symptoms) with a total score range of 0 to 27. Lower scores indicate less depression.
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | 0.0 (0.38) | -0.3 (0.35)

44. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Total Score at Day 5: 70 mg
Description: as for outcome 43
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | -0.4 (0.30) | -0.7 (0.28)

45. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Total Score at Day 5: 100 mg
Description: as for outcome 43
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | -0.4 (0.30) | -0.9 (0.34)

46. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Total Score at Day 5: 150 mg
Description: as for outcome 43
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | -0.7 (0.47) | -1.0 (0.35)

47. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Total Score at Day 5: 200 mg
Description: as for outcome 43
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 22
units on a scale | -0.4 (0.30) | -0.6 (0.28)

48. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Total Score at Day 5: 250 mg
Description: as for outcome 43
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
units on a scale | -0.2 (0.40) | -0.3 (0.48)

49. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at Day 5: 50 mg
Description: SAS is a 10-item scale used to evaluate the presence and severity of extrapyramidal symptoms. The items are scored on a scale from 0 to 4 with item-specific definitions given for each point. Total scores range from 0 to 40. Lower scores indicate less impairment.
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | -0.4 (0.30) | 0.0 (0.18)

50. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at Day 5: 70 mg
Description: as for outcome 49
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | -0.6 (0.43) | -0.1 (0.18)

51. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at Day 5: 100 mg
Description: as for outcome 49
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | -0.4 (0.48) | 0.0 (0.21)

52. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at Day 5: 150 mg
Description: as for outcome 49
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | -0.3 (0.29) | 0.1 (0.19)

53. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at Day 5: 200 mg
Description: as for outcome 49
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 6 | 22
units on a scale | 0.0 (0.52) | 0.0 (0.20)

54. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at Day 5: 250 mg
Description: as for outcome 49
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
units on a scale | 0.2 (0.31) | 0.0 (0.21)

55. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at Day 5: 50 mg
Description: BAS scale has objective, subjective, and global impression components of akathisia (motor restlessness that manifests itself with an inability to sit still or remain motionless). Objective and subjective components are rated on a scale from 0 (normal/absence) to 3 (severe) and are summed yielding a total score of 0 to 9. Global impression is rated on a scale from 0 (absent) to 5 (severe) with a total score ranging from 0 to 5. Lower scores indicate reduced restlessness.
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | 0.0 (0.00) | 0.0 (0.00)

56. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at Day 5: 70 mg
Description: as for outcome 55
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
units on a scale | 0.0 (0.00) | 0.0 (0.00)

57. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at Day 5: 100 mg
Description: as for outcome 55
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | 0.0 (0.00) | 0.0 (0.00)

58. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at Day 5: 150 mg
Description: as for outcome 55
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
units on a scale | 0.0 (0.00) | 0.0 (0.00)

59. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at Day 5: 200 mg
Description: as for outcome 55
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 22
units on a scale | 0.0 (0.00) | 0.2 (0.11)

60. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at Day 5: 250 mg
Description: as for outcome 55
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
units on a scale | 0.0 (0.00) | 0.0 (0.05)

61. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Groton Maze Learning Test, 50 mg
Description: This battery is a series of 4 computerized cognition tests (Groton Maze Learning Test, Detection Task, Identification Task, and One Card Learning Task) designed to measure reaction time, visual learning and reasoning, and problem solving. The entire battery takes approximately 12 minutes to complete. CogState scores are measured on a linear scale (no maximum score). The Groton Maze Learning Test measures total number of errors made in problem solving (lower score = better performance). The Detection Task is measured by speed of performance (lower score = better performance). The Identification Task is measured by speed of performance (lower score = better performance). One Card Learning Task measures the accuracy of performance (higher score = better performance).
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of Errors
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
Number of Errors | -0.9 (8.02) | -8.2 (5.79)

62. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Groton Maze Learning Test, 70 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of Errors
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
Number of Errors | 8.7 (10.77) | -7.3 (6.45)

63. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Groton Maze Learning Test, 100 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of Errors
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
Number of Errors | 0.9 (9.55) | -15.7 (6.57)

64. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Groton Maze Learning Test, 150 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of Errors
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
Number of Errors | 21.1 (28.75) | -11.3 (6.26)

65. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Groton Maze Learning Test, 200 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of Errors
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 22
Number of Errors | -10.3 (6.30) | -16.5 (6.65)

66. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Groton Maze Learning Test, 250 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of Errors
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
Number of Errors | -5.0 (8.74) | -13.2 (5.25)

67. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Detection Task, 50 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
Log10 milliseconds | 0.0 (0.0389) | -0.034 (0.0223)

68. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Detection Task, 70 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
Log10 milliseconds | 0.017 (0.0411) | -0.015 (0.0195)

69. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Detection Task, 100 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
Log10 milliseconds | 0.014 (0.0492) | -0.047 (0.0246)

70. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Detection Task, 150 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
Log10 milliseconds | 0.037 (0.0373) | -0.039 (0.0180)

71. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Detection Task, 200 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 22
Log10 milliseconds | -0.025 (0.0395) | -0.049 (0.0178)

72. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Detection Task, 250 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
Log10 milliseconds | -0.034 (0.0581) | -0.048 (0.0147)

73. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Identification Task, 50 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
Log10 milliseconds | 0.028 (0.0304) | 0.001 (0.0141)

74. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Identification Task, 70 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
Log10 milliseconds | 0.015 (0.0273) | 0.006 (0.0113)

75. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Identification Task, 100 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
Log10 milliseconds | 0.011 (0.0348) | 0.001 (0.0171)

76. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Identification Task, 150 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
Log10 milliseconds | 0.036 (0.0419) | -0.010 (0.0172)

77. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Identification Task, 200 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 22
Log10 milliseconds | 0.044 (0.0397) | -0.014 (0.0157)

78. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: Identification Task, 250 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
Log10 milliseconds | 0.005 (0.0531) | -0.007 (0.0144)

79. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: One Card Learning Task, 50 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Arcsine proportion correct
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg)
Number analyzed (Participants) | 7 | 24
Arcsine proportion correct | 0.025 (0.0234) | 0.005 (0.0179)

80. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: One Card Learning Task, 70 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Arcsine proportion correct
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(70 mg)
Number analyzed (Participants) | 7 | 24
Arcsine proportion correct | 0.015 (0.0322) | 0.021 (0.0189)

81. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: One Card Learning Task, 100 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Arcsine proportion correct
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(100 mg)
Number analyzed (Participants) | 7 | 23
Arcsine proportion correct | 0.012 (0.0373) | 0.012 (0.0197)

82. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: One Card Learning Task, 150 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Arcsine proportion correct
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(150 mg)
Number analyzed (Participants) | 7 | 23
Arcsine proportion correct | 0.026 (0.0415) | 0.042 (0.0222)

83. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: One Card Learning Task, 200 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Arcsine proportion correct
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(200 mg)
Number analyzed (Participants) | 7 | 22
Arcsine proportion correct | -0.020 (0.0394) | 0.046 (0.0219)

84. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at Day 5: One Card Learning Task, 250 mg
Description: as for outcome 61
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Arcsine proportion correct
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(250 mg)
Number analyzed (Participants) | 6 | 22
Arcsine proportion correct | 0.018 (0.0432) | 0.022 (0.0250)

ADVERSE EVENTS:
Groups:
- SPD489 (Lisdexamfetamine Dimesylate)(50 mg); SPD489 (Lisdexamfetamine Dimesylate)(70 mg); SPD489 (Lisdexamfetamine Dimesylate)(100 mg); SPD489 (Lisdexamfetamine Dimesylate)(150 mg); SPD489 (Lisdexamfetamine Dimesylate)(200 mg); SPD489 (Lisdexamfetamine Dimesylate)(250 mg); SPD489 (Lisdexamfetamine Dimesylate)(All Doses): Ascending multiple, oral doses of SPD489 (50mg, 70mg, 100mg, 150mg, 200mg, 250mg) administered once daily for 5 days at each dose level (30 days total).
Arm/Group | Placebo | SPD489 (Lisdexamfetamine Dimesylate)(50 mg) | SPD489 (Lisdexamfetamine Dimesylate)(70 mg) | SPD489 (Lisdexamfetamine Dimesylate)(100 mg) | SPD489 (Lisdexamfetamine Dimesylate)(150 mg) | SPD489 (Lisdexamfetamine Dimesylate)(200 mg) | SPD489 (Lisdexamfetamine Dimesylate)(250 mg) | SPD489 (Lisdexamfetamine Dimesylate)(All Doses)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/24 | 0/24 | 0/24 | 0/23 | 0/23 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 4/7 | 15/24 | 7/24 | 8/24 | 12/23 | 10/23 | 12/22 | 23/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | SPD489 (Lisdexamfetamine Dimesylate)(50 mg) (N=24) | SPD489 (Lisdexamfetamine Dimesylate)(70 mg) (N=24) | SPD489 (Lisdexamfetamine Dimesylate)(100 mg) (N=24) | SPD489 (Lisdexamfetamine Dimesylate)(150 mg) (N=23) | SPD489 (Lisdexamfetamine Dimesylate)(200 mg) (N=23) | SPD489 (Lisdexamfetamine Dimesylate)(250 mg) (N=22) | SPD489 (Lisdexamfetamine Dimesylate)(All Doses) (N=24)
Tachycardia (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 6 (8)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 4 (7)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (8)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 4 (5) | 4 (13)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 5 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Increased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope Vasovagal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.